CLINICAL TRIAL: NCT06606483
Title: A 24 Weeks, Multicenter, Randomized, Double-blind, Placebo, Parallel-controlled Phase IIb Trail Comparing the Efficacy and Safety of MDR-001 Tablet Versus Placebo in Subjects With Overweight or Obesity
Brief Title: A Study to Evaluate the Efficacy and Safety of MDR-001 in Subjects Who Are Obesity or Overweight
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MindRank AI Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MDR-001-CN-02
Record Dates: First submitted 2024-09-16; First posted 2024-09-23 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Obesity; Overweight and Obesity
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 90 mg MDR-001 (Experimental): Drug: MDR-001 Administered orally
  Interventions: Drug: MDR-001
- 120 mg MDR-001 (Experimental): Drug: MDR-001 Administered orally
  Interventions: Drug: MDR-001
- 150 mg MDR-001 (Experimental): Drug: MDR-001 Administered orally
  Interventions: Drug: MDR-001
- 180 mg MDR-001 (Experimental): Drug: MDR-001 Administered orally
  Interventions: Drug: MDR-001
- placebo (Placebo Comparator): Drug: MDR-001 Administered orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MDR-001 — Oral administration of small molecule MDR-001 tablets
  Arms: 120 mg MDR-001; 150 mg MDR-001; 180 mg MDR-001; 90 mg MDR-001
Drug: Placebo — Administered orally placebo
  Arms: placebo

SUMMARY:
This is a 24 weeks, multicenter, randomized, double-blind, placebo, parallel-controlled Phase IIb trail comparing the efficacy and safety of MDR-001 tablet versus placebo as an adjunct to a reduced calorie diet and increased physical activity in subjects with overweight or obesity, and to explore the optimal dose selection to support the subsequent Pivotal trial.

ELIGIBILITY:
Inclusion Criteria:

1. In accordance with adequate informed consent, the subject voluntarily signs the Informed Consent Form (ICF).
2. Male or female participants aged ≥18 and ≤ 65 years, who have signed the Informed Consent Form (ICF)
3. Have BMI of

   • obesity: ≥28 kg/m2
   * overweight: ≥24 kg/m2 and ≤28 kg/m2 with at least 1 of the following weight-related comorbidities

     1) prediabetes: 6.1 mmol/L (110 mg/dL) ≤FPG≤7.0 mmol/L (126 mg/dL) ; and/or 5.7%≤HbA1c≤6.5% 2）Hypertension: medical record for Hypertension, or diagnosis of hypertension for the first time during screening (with at least three measurements spaced across at least over a period of two days, defining hypertension as a systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg).

     3) Dyslipidemia: medical record for dyslipidemia (regardless of medication treatment) or TC≥5.2 mmol/L (200 mg/dl), and/or LDL-C≥3.4 mmol/L (130 mg/dl), and/or HDL-C<1.0 mmol/L (40 mg/d l), and/or TG≥1.7 mmol/L (150 mg/dl) at screening 4) fatty liver disease(FLD): Presence of FLD confirmed by imaging studies within three months prior to screening, or diagnosis of FLD at screening 5) obstructive sleep apnea 6) Presence of weight-bearing joint pain during the screening period or within three months prior to screening. (Acceptance of patient self-description)
4. The weight change achieved through dietary and exercise control should not exceed a 5% variation within three months prior to screening. (Acceptance of patient self-description)
5. Potential participants with fertility potential (including the partners of male participants) must not have any plans for conception or sperm donation from the screening period until 6 months after the last dose administration, and they should be willing to use at least one effective contraception method.
6. The participant must have a thorough understanding of the trial objectives, be able to communicate effectively with the investigators, and be capable of comprehending and adhering to all the requirements of this trial, including following the medication regimen and lifestyle guidance as outlined in the protocol.

Exclusion Criteria:

1. Have obesity induced by other disorders or drugs, including elevated cortisol hormones (such as Cushing's syndrome), polycystic ovary syndrome, obesity due to pituitary and hypothalamic injuries, etc
2. Previous diagnosis of diabetes mellitus (including Type 1 diabetes, Type 2 diabetes, diabetes caused by pancreatic injury, or other types of diabetes) or diagnosis of Type 2 diabetes at the time of screening/randomization, defined as: HbA1c ≥ 6.5%; and/or fasting plasma glucose ≥ 7.0 mmol/L (126 mg/dL); and/or random plasma glucose ≥ 11.1 mmol/L (200 mg/dL).
3. A history of at least one episode of hypoglycemia occurring within the 3 months prior to screening, without apparent precipitating causes, is defined as FPG <2.8 mmol/L (50 mg/dL) and/or the presence of marked symptoms of hypoglycemia.
4. A history of psychiatric disorders, addictive diseases, or other conditions that may impair the ability of the participant to provide informed consent.
5. A history of suicidal ideation or suicidal behavior.
6. Have any of the following major cardiovascular and cerebrovascular conditions within 6 months prior to Screening 1) myocardial infarction(MI), percutaneous coronary intervention(PCI), coronary artery bypass grafting(CABG), heart valve repair/replacement, unstable angina, hemorrhagic stroke (stroke), ischemic stroke (including transient ischemic attack (TIA)); 2) New York Heart Association Functional Classification III or IV congestive heart failure
7. A history of gout within the past six months prior to screening.
8. A history of proliferative retinopathy or macular degeneration.
9. Have a history of malignancy less than 5 years or diagnosis of malignancy at screening (other than cured basal cell skin cancer, or in situ carcinomas of the cervix)
10. Have a known self or family history (first-degree relative) of medullary thyroid carcinoma or multiple endocrine neoplasia type 2
11. Have a personal or family history of long QT syndrome, family history of sudden death in a first-degree relative (parents, siblings, or children) before the age of 40 years, and/or a personal history of unexplained syncope within the last year.
12. During the screening phase, subjects exhibited thyroid function abnormalities uncontrolled (TSH>6 mIU/L or <0.4 mIU/L) by a stable medication regimen (stable dosages for three months or more), Subclinical hypothyroidism requiring no treatment (with TSH levels <10.0 mIU/L and normal range of FT3 and FT4) is excluded.
13. Within the six months preceding screening, subjects experienced severe gastrointestinal disorders (such as active gastric ulcers), or underwent gastrointestinal surgery (Appendectomy, cholecystectomy, or other gastrointestinal endoscopic surgeries deemed by the investigator to have no significant impact on gastrointestinal motility are excluded), or have a known clinically significant gastric emptying abnormality (for example, pyloric obstruction, gastroparesis)
14. Amylase/lipase>3 ULN at screening or have had a history of chronic or acute pancreatitis
15. Have had a history of chronic or acute hepatitis; or have signs and symptoms of any other liver disease other than nonalcoholic fatty liver disease at screening, or any of the following, as determined by the laboratory during screening 1）ALT or AST ≥3×ULN 2）TBIL≥1.5×ULN 3）ALP≥3×ULN
16. Subjects with a history of acute biliary tract disease (cholecystitis, gallstones, or bile duct stones) within one year prior to screening, or suffer from biliary tract disease accompanied by related clinical symptoms which should be treated at screening/randomization, are deemed unsuitable for participation in this clinical trial by the investigator.
17. The subjects exhibit hypersensitivity or a suspected hypersensitivity to GLP-1 receptor agonists (GLP-1RAs) or to excipients.
18. Have a history of drug or alcohol abuse
19. Have a history of alcoholism within the prior 3 months of study screening (750 mL of beer or 250 mL of wine or 50 g of distilled spirits per day)
20. Have taken within 3 months prior to screening medications or food intended to affect body weight, including but not limited to:

1) Approved/unapproved weight-loss drugs: Orlistat, Sibutramine Hydrochloride, Phentermine Resin Complex, Phentermine-Topiramate, Contrave, Semaglutide, Liraglutide, Phendimetrazine, Methamphetamine, etc.; 2) GLP-1RA or GLP-1R/GCGR or GIPR/GLP-1R or GIPR/GLP-1R/GCGR or DPP-4 inhibitors 3) Hypoglycemic drugs, such as metformin, sodium-glucose cotransporter 2 (SGLT2) inhibitors, thiazolidinediones (TZDs), etc.

4) Systemic steroids (including intravenous, oral, intra-articular administration) 5) Tricyclic antidepressants or other antipsychotic or antiepileptic drugs intended to affect body weight (such as: Mirtazapine, Paroxetine, Clozapine, Olanzapine, Risperidone, Paliperidone, Valproic acid, Valproic acid derivatives, lithium salt).

21. Have a prior or planned surgical treatment for obesity (excluding acupuncture, cupping, thread lift, liposuction or abdominoplasty, if performed 1 year prior to screening) or planned surgical treatment or acupuncture, cupping, thread lift, liposuction or abdominoplasty during clinical trial 22. Screening within 3 months before the large or medium-sized surgery or serious trauma, severe infection occurred, the investigator judged not suitable for this trial or during the trial period is planned to receive surgery (Outpatient surgeries that are judged by the investigator to have no impact on the safety of the subjects and the results of the trial are excluded) 23. Have had a history of organ transplantation 24. The use of any drugs or foods known to potently or moderately inhibit CYP3A4 and/or P-gp is prohibited within 28 days prior to the first administration of the study drug and throughout the duration of the trial.

25. Have poorly controlled hypertension (mean seated systolic BP ≥160 mm Hg or mean seated diastolic BP ≥100 mm Hg) at screening (Pre-randomization review; seated, at rest for at least 5 minutes, with a second measurement taken to average the values if the difference between the two measurements exceeds ≥5 mmHg, with a third measurement taken if necessary, with at least a one-minute interval between each test. The final test result is the arithmetic mean of the three test results) 26. positive HBsAg or HCV antibodies or HIV antibodies or syphilis antibodies at screening 27. During the screening phase, laboratory examination results meet any of the following criteria:

1. calcitonin≥50 ng/L
2. estimated eGFR ≤60 mL/min/1.73 m2, calculated by CKD-EPI
3. uncontrolled severe dyslipidemia, with triglyceride (TG) levels ≥ 5.65 mmol/L (500 mg/dL) treated by conventional lipid-lowering medications.
4. INR>1.5×ULN
5. hemoglobin value <110 g/L (females) or <120 g/L (males) 28. Screening for QTcF>450 ms (males) and QTcF>470 ms (females) at rest (at least 5 min, repeat measurement once to obtain the average, with a 2 min ± 60 s interval between the two measurements).

29. Participating in another clinical trial; or, if on treatment with the investigational drug or device, the time since the last dose or cessation of treatment is ≤3 months or 5 half-lives (t1/2) of the investigational drug (whichever is longer) prior to the first day of this trial screening.

30. Have a blood transfusion or severe blood loss ≥500 mL within the prior 3 months of study screening or received blood transfusion before screening 31. Pregnant or lactating females; 32. Parties directly associated with this trial, including but not limited to, the principal investigator(s), staff members of the trial centers, and/or their immediate family members. Immediate family members are defined as spouses, parents, children, or siblings, whether born or legally adopted.

33. Inability to complete the trial for reasons unrelated to the study, or any other condition or prior therapy that would make the participant unsuitable for this study (such as participant refusal to adhere to the prescribed weight-loss medication exclusively during the trial period).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-09-23 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Body Weight From Baseline at Week 24 | Baseline, Week 24

SECONDARY OUTCOMES:
Change in Body Weight (kg) from Baseline at Week 24 | Baseline, Week 24
Percentage of Study Participants Who Achieve ≥5% Body Weight Reduction at Week 24 | Baseline, Week 24
Percentage of Study Participants Who Achieve ≥10% Body Weight Reduction at Week 24 | Baseline, Week 24
Change in BMI (kg/m2) from Baseline at Week 24 | Baseline, Week 24
Change in Waist Circumference from Baseline at Week 24 | Baseline, Week 24
Change in hyperlipidemia (TC, TG, LDL-C, HDL-C, nHDL-C) From Baseline at Week 24 | Baseline, Week 24
Change in Blood Pressure (SBP, DBP) from Baseline at Week 24 | Baseline, Week 24
Change in Blood Glucose (HbA1c, FPG) from baseline at Week 24 | Baseline, Week 24

OTHER OUTCOMES:
To assess safety and tolerability of study interventions | up to 25 weeks
The time-course variation of MDR-001 plasma concentration | up to 25 weeks
MDR-001 Population Pharmacokinetic (PopPK) Analysis | up to 25 weeks
Percentage of Study Participants Who Achieve ≥15% Body Weight Reduction at Week 24 | Baseline, Week 24

CONTACTS AND LOCATIONS:
Locations (19):
- China (19):
  - The Second Hospital Of Anhui Medical University, Hefei, Anhui
  - The People's Hospital of Suancheng City, Xuancheng, Anhui
  - Zibo Central Hospital, Zibo, Anhui
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The Third People's Hospital of Hainan, Haikou, Hainan
  - The Second Hospital Of Hebe Medical University, Shijiazhuang, Hebei
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The first Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang, Henan
  - The First People's Hospital of Chenzhou City, Chenzhou, Hunan
  - Zhuzhou Central Hospital, Zhuzhou, Hunan
  - Second Hospital of Jilin University, Changchun, Jilin
  - Daqing People's Hospital, Daqing, Jilin
  - Panjin Liaoyou Gem Flower Hospital, Panjin, Liaoning
  - The Fifth People's Hospital of Shenyang, Shenyang, Liaoning
  - Central hospital of Jinan, Jinan, Shandong
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Xianyan Hospital of Yanan Univisity, Xianyang, Shanxi
  - Yichang Central People's Hospital, Yichang, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided